CLINICAL TRIAL: NCT07023991
Title: Effect of Adding Dexmedetomidine to Bupivacaine in US- Guided Erector Spinae Plane Block for Post-operative Pain Management in Pediatric Patients Undergoing Lower Abdominal Surgeries
Brief Title: Dexmedetomidine Added to Bupivacaine for ESP Block in Children Undergoing Lower Abdominal Surgeries
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MS113/2025
Record Dates: First submitted 2025-05-22; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-02

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine Group (Active Comparator): Patients in this group will receive an ultrasound-guided erector spinae plane (ESP) block with bupivacaine only.
  Interventions: Drug: Bupivacaine
- Bupivacaine + Dexmedetomidine Group (Experimental): Patients in this group will receive an ultrasound-guided erector spinae plane (ESP) block with a combination of bupivacaine and dexmedetomidine.
  Interventions: Drug: Bupivacaine; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine will be used in an ESP block to provide postoperative analgesia.
  Other Names: Marcaine
Drug: Dexmedetomidine — Dexmedetomidine will be added to bupivacaine in the ESP block to evaluate its effect on duration of postoperative analgesia.
  Other Names: Precedex
  Arms: Bupivacaine + Dexmedetomidine Group

SUMMARY:
This study aims to evaluate the effect of adding dexmedetomidine to bupivacaine in erector spinae plane (ESP) blocks on the duration of postoperative analgesia in pediatric patients undergoing lower abdominal surgery. Effective postoperative pain control in children remains a clinical challenge, and regional anesthesia techniques such as the ESP block have shown promise in improving outcomes.

In this randomized, double-blind clinical trial, pediatric patients scheduled for elective lower abdominal surgeries will be assigned to receive either bupivacaine alone or bupivacaine combined with dexmedetomidine as part of an ultrasound-guided ESP block. The primary outcome is the duration of postoperative analgesia, defined as the time from the block until the first request for rescue analgesia. Secondary outcomes include total analgesic consumption and postoperative pain scores

DETAILED DESCRIPTION:
* Preoperative setting:

  * A careful history taking will be done from the parents of the child for any medical disorder such as congenital coagulation disorders or therapeutic anticoagulants.
  * A complete physical examination of the child will be done, including the central nervous system for signs of mental disturbance, the chest for any deformities or chest infection, the heart for congenital heart disease, and the back for any spinal deformities or infection at the site of injection.
  * Routine preoperative investigations will be done to all patients, including laboratory investigations (complete blood picture, liver and kidney function tests, prothrombin time and partial thromboplastin time) and other as needed by the patient condition.
  * Written informed consent will be obtained from all participants' parents or legal guardian prior to the study.
* Intraoperative setting:

  * All children will be premedicated orally with midazolam (0.05-0.1 mg/kg over 2-3 minutes, maximum 6 mg) 30 minutes prior to surgery. On arrival of the patients to the operative room, routine monitoring with 5-leads electrocardiogram (ECG), non-invasive blood pressure (NIBP) and pulse oximetry will be instituted, then anesthesia will be induced with 8% sevoflurane in 100% oxygen. After an adequate depth of anesthesia is reached, an intravenous access will be placed under aseptic condition, then all patients will receive intravenous (IV) fentanyl (1 µg/kg) and atracurium (0.5 mg/kg), and orotracheal endotracheal intubation will be performed. Anesthesia will be maintained with a mixture of oxygen-air (50% - 50%) and isoflurane

    1. -1.5%). Muscle relaxation will be sustained during the procedure with incremental doses of IV atracurium (0.1 mg/kg) every 25 minutes.

       In group A: US guided ESPB will be performed with aseptic precautions using a (6- 19) MHz linear probe in a sterile cover with sterile jelly (GE LOGIQ 5, USA).
  * Technique of US guided ESPB block: The block will be performed by a trained anesthetist in regional anesthetic techniques while the patient in lateral position, the ultrasound transducers will be placed in a parasagittal plane 2-3 cm away from the midline at the level of first lumbar vertebra (L1) (The L1 level will be identified by counting upwards from the sacrum). Sliding the transducer medially till identifying the transverse process which appear as flat acoustic shadow and after identification of erector spinae muscle (ESM) and transverse process, a 22-gauge 50 mm echogenic block needle (Sono Plex® PAJUNK®, Germany) will be introduced in cranio-caudal direction with in-plane technique and after confirming the position of the tip of the needle over the transverse process with negative aspiration to blood or air, Bupivacaine 0.25% (with a maximum dose 2 mg/kg) plus Dexmedetomidine (0.5µg/kg), putting into consideration that the total volume to be 0.3 ml/kg on each side, will be injected. The spread of local anesthetic in a plane below the erector spinae muscle will be visualized.
  * The skin incision will be made 15 min after the block.
  * Baseline values of heart rate (HR) and mean blood pressure (MAP) will be recorded before skin incision and then recorded at 5, 30, 60 minutes after skin incision and at the end of surgery. Also, patients will be monitored for sign of local anesthetic toxicity.
  * Any complications related to the block given will be recorded including hematoma, intravascular injection, and allergic reactions.
  * If local anesthetic toxicity occurred, cardiovascular and respiratory support and 20% intralipid bolus of 1.5 ml/kg over 2-3 min will be given.

In group B: This group will receive ESPB using Bupivacaine 0.25% (with a maximum dose 2 mg/kg) alone 15 min before skin incision with the same protocol and precautions.

* In both group an increase in heart rate to 20% above the baseline values at any time during the procedure will be defined as insufficient analgesia and fentanyl 0.5 µg/kg will be given and the total amount of intraoperative opioid will be recorded.
* At the end of the surgery Isoflurane will be discontinued and neostigmine 0.05 mg/kg plus atropine 0.02 mg/kg will be administered to reverse the effect of atracurium. After awakening from anesthesia and achieving an appropriate level of consciousness, the patient will be discharged from the operating room to be transferred to the PACU (Post Anesthesia Care Unit), and pain assessment will be done immediate post extubating.

Postoperative setting:

* Postoperative pain score will be assessed using FLACC scale immediately after transfer to the PACU, at 1, 2, 4, 6, 8, 12 hours postoperatively and before discharge from hospital.
* If the FLACC score was ≥ 4, analgesia in the form of Paracetamol 15 mg/kg IV will be administered as the first rescue analgesia. The time for the first rescue analgesic administration will be recorded. If this analgesia will not be adequate, intravenous pethidine at 1mg/kg will be given as the second rescue analgesia and the total analgesic requirements of paracetamol and pethidine will be recorded.
* FLACC is a behavioral pain assessment scale used for nonverbal or preverbal patients who are unable to self-report their level of pain. Pain is assessed through observation of five categories including face, legs, activity, cry, and concealability.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients aging 1-7 years old of both sexes.
2. Patients scheduled for unilateral or bilateral lower abdominal surgeries.
3. American Society of Anesthesiologists (ASA) Physical Status Class I, II

Exclusion Criteria:

1. Parents or legal guardian refusal of participation in the study.
2. Contraindication to regional anesthesia (including coagulopathy and local infection).
3. History or known allergy to local anesthetics.
4. Past history of any complications related to the block. (including hematoma and intravascular injection)
5. Spinal anomalies altered mental status, a history of developmental delay.
6. Additional surgical procedures at different surgical sites.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Duration of Postoperative Analgesia | Up to 24 hours after surgery
  Measurement of the time from recovery of anesthesia to the need of first given dose of rescue analgesia.

SECONDARY OUTCOMES:
Postoperative Pain Scores | At 1, 2, 4, 6, 12, and 24 hours after surgery
  * Measured using the Face, Legs, Activity, Cry, Consolability (FLACC) scale.
  * Score range: 0 (no pain) to 10 (severe pain).
  * Higher scores indicate worse pain.
Total intraoperative analgesics | During the operation from the induction of anesthesia until the recovery.
  Total intraoperative fentanyl consumption in micrograms
Total Postoperative Analgesic Consumption | Within 24 hours postoperatively
  The total amount (in milligrams) of rescue analgesics administered to the patient within the first 24 hours after surgery.
Incidence of Adverse Effects | Within 24 hours postoperatively
  The occurrence of adverse effects such as sedation, nausea, vomiting, bradycardia, or hypotension within 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed G Nowar, MBBCH, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once study is completing
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before 1/2026
Access Criteria: Free